CLINICAL TRIAL: NCT01856322
Title: Phase 2 Prospective Randomized Double Blind Trial Comparing Metastasectomy Plus Sulindac Versus Metastasectomy Alone in Patients With Stage IV Colorectal Cancer
Brief Title: Surgery Plus Sulindac or Surgery Alone for Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was prematurely closed due to lack of accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Marybeth Hughes, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130126; 13-C-0126
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer; Liver Metastasis; Colorectal Adenocarcinoma
Keywords: Colorectal Cancer; Liver Metastasis; Sulindac
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sulindac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sulindac (Active Comparator): one tablet twice daily
  Interventions: Drug: Sulindac
- Placebo (Placebo Comparator): one tablet twice daily
  Interventions: Drug: Placebo
- Normal Volunteers (or control group) (Other): Normal volunteers (or control group) enrolled with the only purpose to validate assays and the shipping method.
  Interventions: Other: Validate assays and shipping methods

INTERVENTIONS:
Drug: Sulindac — one tablet 150mg twice daily
  Arms: Sulindac
Drug: Placebo — One tablet twice daily
  Arms: Placebo
Other: Validate assays and shipping methods
  Arms: Normal Volunteers (or control group)

SUMMARY:
Background:

- Some types of inflammation may increase the risk of cancers in the intestinal track. Because of this possibility, anti-inflammatory drugs may be able to prevent tumor growth and spread. One such drug, sulindac, may be helpful to study. Researchers want to see if people who are having surgery to remove intestinal tumors from advanced colorectal cancer will benefit from sulindac. It will be tested against a placebo.

Objectives:

- To see if sulindac can improve treatment outcomes in people who are having surgery for advanced colorectal cancer.

Eligibility:

- Individuals at least 18 years of age who are having surgery for advanced colorectal cancer.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected. Imaging studies and heart and lung function tests may also be given.
* Participants will be separated into two groups. One group will take sulindac. The other will take a placebo.
* Participants will take sulindac or placebo twice daily from about 2 to 3 weeks before the scheduled surgery. Seven days before the surgery, they will stop taking the pills.
* Participants will have surgery to remove their tumors. The surgery will also remove affected organ tissue.
* Participants will start to take the pills again once they have recovered from surgery. They will continue taking the sulindac or placebo twice a day for 3 years, or for as long as the tumors do not return.

DETAILED DESCRIPTION:
* Despite strong evidence for a causative role of inflammatory mediators in intestinal cancer, the underlying mechanisms remain obscure. Established evidence indicates activation of the Wnt/beta-catenin pathway is an early step in the malignant transformation of colorectal adenomas with persistent activation in 90% of colorectal cancers. Activation of this pathway ultimately effects transcription of the S100A4 gene.
* S100A4 transcript serum levels have been shown to correlate with risk of recurrence in colorectal cancer and patients with systemic metastases are found to have increased S100A4 transcript expression.
* S100A4 may be a novel prognostic biomarker in colorectal cancer.
* Cyclooxygenase-2 is a key enzyme involved in the inflammatory response and is a key target of molecular chemoprevention in colorectal adenoma prevention trials.
* Recent studies demonstrate mitigation of Wnt/beta-catenin signaling by COX-2 inhibition via administration of the non-steroidal anti-inflammatory drug (NSAID) sulindac using in vitro and in vivo animal models.
* We hypothesize that sulindac administration will abrogate Wnt/beta-catenin mediated signaling and thus decrease S100A4 activity in patients with colorectal metastases.
* We propose to define the benefit of sulindac administration to patients with colorectal metastases following resection and validate the use of circulating S100A4 transcripts as a novel biomarker for disease recurrence.

ELIGIBILITY:
-INCLUSION CRITERIA

1. Histologically confirmed colorectal adenocarcinoma with metastatic disease confined to the liver, or limited extrahepatic intra-abdominal disease Note: limited sites of disease include:

   * porta hepatis lymph node metastases
   * pelvic lymph node metastases (internal iliac, external iliac or obturator)
2. Hepatic and intra-abdominal metastases must be measurable by computed tomography (CT), magnetic resonance imaging (MRI) and/or positron emission tomography (PET) scan
3. Liver disease must be amenable to gross total resection (R0/R1) with adequate functional liver remnant which requires preservation of at least 2 contiguous hepatic segments with adequate inflow, outflow, and biliary drainage with a functional liver remnant (FLR) volume of more than 20% (for healthy liver)
4. Greater than or equal to 18 years of age.
5. Must be able to understand and sign the Informed Consent Documentation.
6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) less than or equal to 2.
7. Life expectancy of greater than six months.
8. Patients of both genders must be willing to practice birth control during and for one week after taking sulindac/placebo.
9. Hematology:

   * Absolute neutrophil count greater than 1500/mm^3 without the support of Filgrastim.
   * Platelet count greater than 75,000/mm^3.
   * Hemoglobin greater than 8.0 g/dl.
10. Chemistry:

    * Serum creatinine less than or equal to 1.5 mg/dl unless the measured creatinine clearance is greater than 60mL/min/1.73m^2.
    * Total bilirubin less than or equal to 2 mg/dl, except for patients with diagnosis of Gilberts disease or hepatic pedicle obstruction then total bilirubin must be less than or equal to 5 mg/dl.
11. International normalized ratio (INR) less than or equal to 1.8.

INCLUSION CRITERIA for NORMAL VOLUNTEERS

* Age greater than 18
* Able to read and understand the informed consent
* No self-reported co morbidities of history of cancer

EXCLUSION CRITERIA

1. Women of child-bearing potential who are pregnant or breast feeding because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
2. Active systemic infections, coagulation disorders or other major medical illnesses precluding major surgery.
3. Patients receiving warfarin anticoagulation, who cannot be transferred to other agents, such as low molecular weight heparins, anti-factor Xa (anti-Xa) agents, etc.
4. Active bleeding disorders
5. Patients with uncontrolled hypertension (would suggest: systolic blood pressure (SBP)> 155, diastolic blood pressure (DBP)> 90), unstable coronary disease (unstable angina, evidence of congestive heart failure (CHF), or myocardial infarction (MI) within 6-12 months of study)
6. Childs B or C cirrhosis or with evidence of severe portal hypertension by history, endoscopy, or radiologic studies or with evidence of moderate to severe ascites.
7. Prior history of gastrointestinal (GI) bleeding unrelated to a cancer diagnosis

   Note: Patients who have a normal upper and lower endoscopy may be enrolled at the discretion of the principal investigator (PI).
8. Renal insufficiency Discretion of principle investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marybeth S Hughes, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics for Hispanics/Latinos, 2012. CA Cancer J Clin. 2012 Sep-Oct;62(5):283-98. doi: 10.3322/caac.21153. PMID 22987332
- [Background] Obrand DI, Gordon PH. Incidence and patterns of recurrence following curative resection for colorectal carcinoma. Dis Colon Rectum. 1997 Jan;40(1):15-24. doi: 10.1007/BF02055676. PMID 9102255
- [Background] de Gramont A, Figer A, Seymour M, Homerin M, Hmissi A, Cassidy J, Boni C, Cortes-Funes H, Cervantes A, Freyer G, Papamichael D, Le Bail N, Louvet C, Hendler D, de Braud F, Wilson C, Morvan F, Bonetti A. Leucovorin and fluorouracil with or without oxaliplatin as first-line treatment in advanced colorectal cancer. J Clin Oncol. 2000 Aug;18(16):2938-47. doi: 10.1200/JCO.2000.18.16.2938. PMID 10944126

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The normal volunteer (or control group) was not randomized to receive medication and was not considered evaluable. The control group purpose is to validate the assays and the shipping methods.
Groups:
- Sulindac: one tablet twice daily
  Sulindac: one tablet twice daily
Period: Overall Study
Arm/Group | Sulindac | Placebo | Normal Volunteers (or Control Group)
Started | 0 | 0 | 3
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 3
Not completed — off study due to lack of accrual | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulindac | Placebo | Normal Volunteers (or Control Group) | Total
Number analyzed (Participants) | 0 | 0 | 3 | 3
Age, Categorical [Number; unit: participants]
  <=18 years |  |  | 0 | 0
  Between 18 and 65 years |  |  | 3 | 3
  >=65 years |  |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 72 (0) | 72 (0)
Gender [Number; unit: participants]
  Female |  |  | 1 | 1
  Male |  |  | 2 | 2
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino |  |  | 0 | 0
  Not Hispanic or Latino |  |  | 3 | 3
  Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native |  |  | 0 | 0
  Asian |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
  Black or African American |  |  | 2 | 2
  White |  |  | 1 | 1
  More than one race |  |  | 0 | 0
  Unknown or Not Reported |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Difference in Circulating S100A4 Transcript in Patients Receiving Sulindac 150 mg BD (Twice Daily) by Mouth Following Resection of Colorectal Cancer Metastases Compared to Those Who do Not.
Description: Difference in circulating S100A4 transcript levels will be determined by assessing the circulating S100A4 transcript level at initial presentation versus the circulating S100A4 transcript level post resection.
Time Frame: 3 years
Population: The trial was prematurely closed due to lack of accrual, thus the outcome measure was not met.
Arm/Group | Sulindac | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sulindac | Placebo | Normal Volunteers (or Control Group)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No